CLINICAL TRIAL: NCT01747252
Title: Randomized Three-way Cross-over Comparative Pharmacokinetic Study of Resveratrol Comprising Products in Fasting Healthy Subjects
Brief Title: Pharmacokinetics of Resveratrol Comprising Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fruitura Bioscience Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 08/12
Record Dates: First submitted 2012-12-09; First posted 2012-12-11 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
MeSH Terms: interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- RGC1 (Experimental): RGC containing the equivalent of 50 mg resveratrol
  Interventions: Dietary Supplement: RGC
- Resveratrol (Active Comparator): The equivalent of 150 mg resveratrol
  Interventions: Dietary Supplement: Resveratrol
- RGC2 (Experimental): RGC containing the equivalent of 150 mg resveratrol
  Interventions: Dietary Supplement: RGC

INTERVENTIONS:
Dietary Supplement: RGC
  Arms: RGC1
Dietary Supplement: RGC
  Arms: RGC2
Dietary Supplement: Resveratrol — The equivalent of 150 mg resveratrol
  Other Names: Transmax (Biotivia Ltd.)
  Arms: Resveratrol

SUMMARY:
This study was designed to assess the pharmacokinetics of 2 doses of Red Grape Cells (RGC) containing resveratrol compared with a reference. RGC will be administered as single oral dose to fasting healthy volunteers. Plasma concentration of free resveratrol and total conjugates will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-55 years;
* BMI >/= 19 and </= 30
* non smoking
* without history or evidence of significant cardiovascular, hepatic, renal, respiratory, gastrointestinal disease
* normal physical and laboratory examinations

Exclusion Criteria:

* History or evidence of alcohol or drug abuse
* subjects receiving chronic medication
* unusual dietary habits or a recent change in body weight
* acute medical situation 48 hours prior to initiation of the study
* poor venous access
* Subjects participated in a trial or donated blood within 4 weeks before initiation of the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Individual plasma concentrations of free and conjugated resveratrol | 24 hours
  Pharmacokinetic data such as the peak plasma concentration (Cmax), time to peak (Tmax) ans area under the concentration-time curves (AUCt) will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- BioStudies Center, Beersheba, Israel

REFERENCES:
- [Derived] Azachi M, Yatuv R, Katz A, Hagay Y, Danon A. A novel red grape cells complex: health effects and bioavailability of natural resveratrol. Int J Food Sci Nutr. 2014 Nov;65(7):848-55. doi: 10.3109/09637486.2014.917152. Epub 2014 May 15. PMID 24827888